CLINICAL TRIAL: NCT02490020
Title: A Perspective Multicenter Controlled Study On Application Of Mesenchymal Stem Cell(MSC) To Prevent Rejection After Renal Transplantation By Donation After Cardiac Death
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Qipeng Sun (Other)
Collaborators: Zhujiang Hospital (Other); The Second Affiliated Hospital, Guangzhou University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor-Investigator, Qipeng Sun, MD, Third Affiliated Hospital, Sun Yat-Sen University
Organization: Third Affiliated Hospital, Sun Yat-Sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: zssy20150624
Record Dates: First submitted 2015-06-29; First posted 2015-07-03 (Estimated); Last update posted 2015-07-03 (Estimated); Status verified 2015-07

CONDITIONS: Disorder Related to Renal Transplantation; Renal Transplant Rejection
Keywords: Renal transplantation; mesenchymal stem cell; Transplantation Rejection; donation after cardiac death

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (8):
- iv of BMSC to prevent rejection (Experimental): Routine treatment protocol(ATG 50mg*3;MP 2.0g to Pred 30mg,then maintaining 5mg qd;MMF 1.0 bid from the first day after op,then maintaining 1-1.5g/d;Plus CNI from the third day after op)+BMSC iv(2*10^6cell/kg, 48h before op)
  Interventions: Biological: mesenchymal stem cell
- routine treatment protocol to prevent rejection (No Intervention): Routine treatment protocol(ATG 50mg*3;MP 2.0g to Pred 30mg,then maintaining 5mg qd;MMF 1.0 bid from the first day after op,then maintaining 1-1.5g/d;Plus CNI from the third day after op)
- ia and iv of MSC to prevent rejection (Experimental): Routine treatment protocol(ATG 50mg*3;MP 2.0g to Pred 30mg,then maintaining 5mg qd;MMF 1.0 bid from the first day after op,then maintaining 1-1.5g/d;Plus CNI from the third day after op)+BMSC (iv 2*10^6cell/kg + ia 5*10^6cell, 48h before op)
  Interventions: Biological: mesenchymal stem cell
- routine treatment to prevent rejection (No Intervention): Routine treatment protocol(ATG 50mg*3;MP 2.0g to Pred 30mg,then maintaining 5mg qd;MMF 1.0 bid from the first day after op,then maintaining 1-1.5g/d;Plus CNI from the third day after op)
- Routine CMR treatment plus MSC to prevent CMR (Experimental): Routine CMR treatment protocol(MP as first line approach, ATG as second line approach,ATG be used to treat BPAR in 1 week after op)+MSC( iv 2*10^6cell/kg at d1,d7)
  Interventions: Biological: mesenchymal stem cell
- Routine CMR treatment to prevent CMR (No Intervention): Routine CMR treatment protocol(MP as first line approach, ATG as second line approach,ATG be used to treat BPAR in 1 week after op)
- Routine AMR treatment plus MSC to prevent AMR (Experimental): Routine AMR treatment protocol(plasma exchange and IVIG as first line approach, anti-CD20 monoclonal antibody as second line approach)+MSC( iv 2*10^6cell/kg at d1,d7)
  Interventions: Biological: mesenchymal stem cell
- Routine AMR treatment to prevent AMR (No Intervention): Routine AMR treatment protocol(plasma exchange and IVIG as first line approach, anti-CD20 monoclonal antibody as second line approach)

INTERVENTIONS:
Biological: mesenchymal stem cell
  Arms: Routine AMR treatment plus MSC to prevent AMR; Routine CMR treatment plus MSC to prevent CMR; ia and iv of MSC to prevent rejection; iv of BMSC to prevent rejection

SUMMARY:
Although donation after cardiac death(DCD) is the major source of renal transplantation in China, high incidence rate of rejection and delayed graft function(DGF) is existing due to the prolonged ischemia time. According to the previous single center study, mesenchymal stem cell (MSC) had an effect to prevent rejection and DGF after renal transplantation, but there was no perspective multicenter controlled study to confirm it. This perspective multicenter controlled study will focus on clarifying the key role of MSC applied via renal arterial or peripheral vein injection, to reduce the rejection and DGF after renal transplantation. The investigators have established GMP workshop and solid research foundation of transplant rejection. This study will provide a new reasonable way for immune induction of renal transplantation by DCD.

ELIGIBILITY:
Inclusion Criteria:

1. Study on prevention of MSC to rejection after transplantation

   * Age between 18-60 years
   * having the indication of renal transplantation
   * having no absolute contraindication
   * renal transplantation by donation after citizen death
   * the first time to receive renal transplantation
   * signed informed consent
2. Study on treatment of MSC to rejection after transplantation

   * renal transplantation by donation after citizen death
   * BPAR
   * having no contraindication of renal biopsy
   * signed informed consent

Exclusion Criteria:

* loss to follow-up
* serious adverse events

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 260 (Estimated)
Dates: Start 2016-01; Primary Completion 2016-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Numbers of participants enrolled into the MSC group and control group | up to one year
  80-100 cases will be enrolled to the group.
Incident rates of BPAR and DGF after renal transplantation with MSC prevention before operation | up to one year
  Cases enrolled into the group will be monitored renal function,renal biopsy and other opportunistic infection.The incident rates of DGF and BPAR will be calculated and compare with the control group.

CONTACTS AND LOCATIONS:
Overall Officials: Qiquan Sun, MD,PhD, Study Director — Third Affiliated Hospital, Sun Yat-Sen University

REFERENCES:
- [Derived] Sun Q, Huang Z, Han F, Zhao M, Cao R, Zhao D, Hong L, Na N, Li H, Miao B, Hu J, Meng F, Peng Y, Sun Q. Allogeneic mesenchymal stem cells as induction therapy are safe and feasible in renal allografts: pilot results of a multicenter randomized controlled trial. J Transl Med. 2018 Mar 7;16(1):52. doi: 10.1186/s12967-018-1422-x. PMID 29514693
- [Derived] Sun Q, Hong L, Huang Z, Na N, Hua X, Peng Y, Zhao M, Cao R, Sun Q. Allogeneic mesenchymal stem cell as induction therapy to prevent both delayed graft function and acute rejection in deceased donor renal transplantation: study protocol for a randomized controlled trial. Trials. 2017 Nov 16;18(1):545. doi: 10.1186/s13063-017-2291-y. PMID 29145879